CLINICAL TRIAL: NCT05093933
Title: A Pivotal Phase 3 Randomized, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of the sGC Stimulator Vericiguat/MK-1242 in Adults With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: A Study of Vericiguat (MK-1242) in Participants With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF) (MK-1242-035)
Acronym: VICTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1242-035; MK-1242-035 (Other: MSD); 2022-500881-80-00 (Registry Identifier: EU CT); U1111-1278-5066 (Registry Identifier: UTN); 2020-005941-18 (EudraCT Number)
Record Dates: First submitted 2021-10-18; First posted 2021-10-26 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vericiguat (Experimental): Participants receive a starting dose of 2.5 mg of vericiguat taken orally once daily. The vericiguat dose will be titrated to 5 mg and to 10 mg.
  Interventions: Drug: Vericiguat
- Placebo (Placebo Comparator): Participants receive a starting matching placebo to vericiguat dose of 2.5 mg taken orally once daily. The matching placebo dose will be sham titrated to 5 mg and to 10 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat — 2.5, 5.0, or 10.0 mg orally once daily
  Other Names: MK-1242; BAY 1021189
  Arms: Vericiguat
Drug: Placebo — 0 mg matching placebo for 2.5 mg, 5 mg, and 10 mg of vericiguat
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vericiguat in participants with chronic heart failure with reduced ejection fraction (HFrEF), specifically those with symptomatic chronic HFrEF who have not had a recent hospitalization for heart failure or need for outpatient intravenous (IV) diuretics. The primary hypothesis is that vericiguat is superior to placebo in reducing the risk of cardiovascular death or heart failure hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic HF [New York Heart Association (NYHA) Class II to IV] on guideline-directed medical therapy for heart failure (GDMT) with no HF hospitalization within 6 months or outpatient IV diuretic use within 3 months before randomization.
* Left ventricular ejection fraction (LVEF) of ≤40%, assessed within 12 months before randomization by any imaging method.
* Elevated N-terminal pro-brain natriuretic peptide (NT-proBNP) levels.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP), or is a WOCBP and agrees to follow contraceptive guidance during the study intervention period and for at least 1 month after the last dose of study intervention.

Exclusion Criteria:

* Has SBP <100 mm Hg or symptomatic hypotension.
* Awaiting heart transplantation, is receiving continuous IV infusion of an inotrope, or has or anticipates receiving an implanted ventricular assist device.
* Amyloidosis or sarcoidosis.
* Primary valvular heart disease requiring surgical procedure or intervention or has undergone a valvular surgical procedure or intervention within 3 months before randomization.
* Hypertrophic cardiomyopathy.
* Acute myocarditis or Takotsubo cardiomyopathy.
* History of heart transplant.
* Tachycardia-induced cardiomyopathy and/or uncontrolled tachyarrhythmia.
* Acute coronary syndrome, or undergone coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within 3 months before randomization.
* History of symptomatic carotid stenosis, transient ischemic attack (TIA), or stroke within 3 months before randomization.
* Malignancy or other noncardiac condition limiting life expectancy to <3 years.
* Requires continuous home oxygen for severe pulmonary disease.
* Interstitial lung disease.
* Discontinuation or dose modification of GDMT or vericiguat within 4 weeks before randomization.
* Recent history (within the last year) of drug or alcohol abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6106 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (519):
- United States (84):
  - Advanced Cardiovascular - Alexander City ( Site 0038), Alexander City, Alabama
  - University of Alabama at Birmingham - School of Medicine-Cardiology ( Site 0153), Birmingham, Alabama
  - Heart Center Research, LLC ( Site 0156), Huntsville, Alabama
  - Mercy Gilbert Medical Center-Dignity Health Cardiology ( Site 0075), Gilbert, Arizona
  - Valley Clinical Trials, Inc. ( Site 0085), Covina, California
  - VA West Los Angeles Medical Center-Cardiology ( Site 0149), Los Angeles, California
  - Valley Clinical Trials Inc ( Site 0006), Northridge, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center ( Site 0010), Torrance, California
  - Blue Coast Research Center ( Site 0053), Vista, California
  - Excel Medical Clinical Trials ( Site 0008), Boca Raton, Florida
  - Universal Axon Clinical Research, LLC ( Site 0022), Doral, Florida
  - Holy Cross Hospital ( Site 0100), Fort Lauderdale, Florida
  - Indago Research and Health Center Inc ( Site 0011), Hialeah, Florida
  - South Florida Research Solutions ( Site 0058), Hollywood, Florida
  - University of Florida - Jacksonville ( Site 0169), Jacksonville, Florida
  - East Coast Institute for Research, LLC ( Site 0047), Jacksonville, Florida
  - Cardiovascular Research Center of South Florida ( Site 0074), Miami, Florida
  - ProLive Medical Research ( Site 0032), Miami, Florida
  - Peace River Cardiovascular Center ( Site 0088), Port Charlotte, Florida
  - BAYCARE MEDICAL GROUP ( Site 0099), Safety Harbor, Florida
  - East Coast Institute for Research - St. Augustine ( Site 0016), Saint Augustine, Florida
  - Cardiovascular Center of Sarasota ( Site 0154), Sarasota, Florida
  - Emory University School of Medicine ( Site 0123), Atlanta, Georgia
  - IACT Health ( Site 0106), Columbus, Georgia
  - NSC Research ( Site 0068), Johns Creek, Georgia
  - Georgia Arrhythmia Consultants and Research Institute ( Site 0042), Macon, Georgia
  - Cardiovascular Consultants of South Georgia, LLC ( Site 0137), Thomasville, Georgia
  - Mount Sinai Hospital ( Site 0050), Chicago, Illinois
  - Chicago Medical Research ( Site 0086), Hazel Crest, Illinois
  - OSF Healthcare Cardiovascular Institute ( Site 0122), Peoria, Illinois
  - Methodist Medical Center of Illinois ( Site 0098), Peoria, Illinois
  - Franciscan Physician Network - Indiana Heart Physicians ( Site 0087), Indianapolis, Indiana
  - The Heart Center of Lake County Research Institute-Research ( Site 0147), Merrillville, Indiana
  - Cardiovascular Research of Northwest Indiana ( Site 0036), Munster, Indiana
  - Reid Physician Associates ( Site 0054), Richmond, Indiana
  - University of Iowa ( Site 0005), Iowa City, Iowa
  - Alliance for Multispecialty Research, LLC ( Site 0143), Wichita, Kansas
  - Norton Healthcare-Norton Heart Specialist ( Site 0062), Louisville, Kentucky
  - Cambridge Medical Trials ( Site 0041), Alexandria, Louisiana
  - Louisiana Heart Center - Hammond ( Site 0004), Hammond, Louisiana
  - The Heart Clinic - Hammond ( Site 0155), Hammond, Louisiana
  - Cardiovascular Institute of the South ( Site 0072), Houma, Louisiana
  - Cardiovascular Institute of the South, 3 ( Site 0096), Lafayette, Louisiana
  - IMA Clinical Research ( Site 0112), Monroe, Louisiana
  - Cardiovascular Institute of the South ( Site 0081), Opelousas, Louisiana
  - Maryland Cardiovascular Specialists ( Site 0056), Baltimore, Maryland
  - Capitol Cardiology Associates - Lanham Office-Maryland Research Centers ( Site 0167), Lanham, Maryland
  - Ascension Providence Hospital ( Site 0094), Southfield, Michigan
  - Phillips Medical Services ( Site 0070), Jackson, Mississippi
  - The University of Mississippi Medical Center-Cardiovascular ( Site 0073), Jackson, Mississippi
  - University of Missouri Hospital ( Site 0163), Columbia, Missouri
  - Washington University-Department of Medicine ( Site 0044), St Louis, Missouri
  - St. Louis Heart and Vascular, P.C.-Clinical Trials Unit ( Site 0029), St Louis, Missouri
  - Logan Health Research ( Site 0017), Kalispell, Montana
  - Renown Regional Medical Center-Renown Institute for Heart and Vascular Health ( Site 0168), Reno, Nevada
  - Amici Clinical Research LLC-Research ( Site 0037), Raritan, New Jersey
  - The Valley Hospital ( Site 0035), Ridgewood, New Jersey
  - Cardiovascular Associates of the Delaware Valley ( Site 0097), Washington Township, New Jersey
  - Erie County Medical Center ( Site 0160), Buffalo, New York
  - New York Presbyterian Medical Group Hudson Valley Cardiology ( Site 0127), Cortlandt Manor, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0161), New York, New York
  - CHEAR Center LLC ( Site 0009), The Bronx, New York
  - Southeastern Cardiology and Cardiovascular-Duke HC CRU - Lumberton ( Site 0134), Lumberton, North Carolina
  - Accellacare - Wilmington ( Site 0090), Wilmington, North Carolina
  - Aultman Hospital-Cardiology Clinical Trials ( Site 0064), Canton, Ohio
  - University of Cincinnati Medical Center-Cardiology ( Site 0071), Cincinnati, Ohio
  - ProMedica Toledo Hospital-ProMedica Heart Failure Clinic ( Site 0061), Toledo, Ohio
  - Doylestown Hospital-Cardiology ( Site 0030), Doylestown, Pennsylvania
  - Accellacare - Charleston ( Site 0141), Charleston, South Carolina
  - Apex Research Foundation ( Site 0001), Jackson, Tennessee
  - Vanderbilt University Medical Center-Vanderbilt Heart and Vascular Institue ( Site 0060), Nashville, Tennessee
  - Dallas VA Medical Center ( Site 0084), Dallas, Texas
  - Southwest Family Medicine Associates ( Site 0131), Dallas, Texas
  - Medresearch Inc ( Site 0043), El Paso, Texas
  - West Houston Area Clinical Trial Consultants ( Site 0014), Houston, Texas
  - South Texas Cardiovascular Consultants, PLLC-Research ( Site 0024), Kerrville, Texas
  - South Texas Cardiovascular Consultants, PLLC-Research ( Site 0020), San Antonio, Texas
  - Tyler Cardiovascular Consultants ( Site 0039), Tyler, Texas
  - INOVA Fairfax Medical Campus ( Site 0136), Falls Church, Virginia
  - Carient Heart & Vascular - Manassas ( Site 0059), Manassas, Virginia
  - Sentara Norfolk General Hospital ( Site 0114), Norfolk, Virginia
  - Dominion Medical Associates, Inc. ( Site 0089), Richmond, Virginia
  - Pulse Heart Institute - Puyallup ( Site 0119), Puyallup, Washington
  - MultiCare Health System-MultiCare Cardiology - Inland Northwest ( Site 0102), Spokane, Washington
- Argentina (7):
  - CEDIC ( Site 4363), CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME)-Cardiology ( Site 4352), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - DIM Clínica Privada ( Site 4359), Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate ( Site 4360), Zárate, Buenos Aires
  - Centro Médico Viamonte-Clinical Research ( Site 4361), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 4356), Rosario, Santa Fe Province
  - Centro de Investigaciones Clinicas del Litoral ( Site 4354), Santa Fe
- Australia (6):
  - Royal Brisbane and Women's Hospital-Cardiology Research ( Site 0453), Brisbane, Queensland
  - The Prince Charles Hospital-Cardiology Research Centre ( Site 0451), Brisbane, Queensland
  - Core Research Group ( Site 0452), Brisbane, Queensland
  - Royal Adelaide Hospital-Cardiology ( Site 0456), Adelaide, South Australia
  - Flinders Medical Centre-Cardiology Research ( Site 0455), Bedford Park, South Australia
  - St. John of God Subiaco Hospital ( Site 0457), Subiaco, Western Australia
- Austria (5):
  - Medizinische Universität Graz-Department of Cardiology ( Site 0351), Graz, Styria
  - Krankenhaus St. Josef Braunau ( Site 0354), Braunau am Inn, Upper Austria
  - Imed19-privat ( Site 0353), Vienna, Vienna
  - Uniklinikum Salzburg-Universitätsklinik für Innere Medizin II, Kardiologie, Internistische Intensiv, Salzburg
  - Klinik Floridsdorf-Karl Landsteiner Institute for Cardiovascular and Critical Care Research c/o Dep, Vienna
- Brazil (10):
  - Hospital de Messejana Dr Carlos Alberto Studart Gomes ( Site 0560), Fortaleza, Ceará
  - Universidade Federal de Goias-Serviço de Cardiologia ( Site 0553), Goiânia, Goiás
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR ( Site 0555), Curitiba, Paraná
  - Hospital Mae de Deus ( Site 0564), Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clinica do Coracao ( Site 0561), Acaraju, Sergipe
  - Instituto de Pesquisa clinica de Campinas ( Site 0551), Campinas, São Paulo
  - CAPED Centro Avancado Pesquisa e Diagnostica ( Site 0552), Ribeirão Preto, São Paulo
  - Hospital de Clínicas de Ribeirão Preto ( Site 0559), Ribeirão Preto, São Paulo
  - Hospital Pro-Cardiaco ( Site 0556), Rio de Janeiro
  - Incor - Instituto do Coracao ( Site 0557), São Paulo
- Canada (21):
  - Heritage Medical Research Clinic ( Site 0679), Calgary, Alberta
  - University Of Alberta Hospital ( Site 0669), Edmonton, Alberta
  - Victoria Heart Institute Foundation ( Site 0680), Victoria, British Columbia
  - St. Boniface General Hospital ( Site 0667), Winnipeg, Manitoba
  - G A Research Associates ( Site 0652), Moncton, New Brunswick
  - NSHA-QEII Health Sciences Centre-Dickson Bldg-Cardiology ( Site 0664), Halifax, Nova Scotia
  - Cambridge Cardiac Care Centre ( Site 0658), Cambridge, Ontario
  - PACE Cardiology ( Site 0675), Newmarket, Ontario
  - North York Diagnostic and Cardiac Centre ( Site 0682), North York, Ontario
  - Oakville Cardiovascular Research LP ( Site 0657), Oakville, Ontario
  - Private Practice - Dr. James Cha ( Site 0655), Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials ( Site 0654), Peterborough, Ontario
  - Corcare-Corcare Cardiovascular Research ( Site 0660), Toronto, Ontario
  - Medicus MFC Research Clinic ( Site 0676), Toronto, Ontario
  - Hôpital de la Cité-de-la-Santé ( Site 0673), Laval, Quebec
  - Institut de Cardiologie de Montreal ( Site 0661), Montreal, Quebec
  - Montreal General Hospital ( Site 0653), Montreal, Quebec
  - Unité de Recherche Clinique du CISSS des Laurentides ( Site 0668), Saint-Jérôme, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer, Sherbrooke, Quebec
  - Hopital Pierre-Le Gardeur ( Site 0674), Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0677), Trois-Rivières, Quebec
- Chile (12):
  - IC La Serena Research ( Site 0769), La Serena, Coquimbo Region
  - Clinica Alemana Osorno ( Site 0768), Osorno, Los Lagos Region
  - Clinical Research Chile SpA ( Site 0761), Valdivia, Los Ríos Region
  - Enroll SpA ( Site 0755), Santiago, Region M. de Santiago
  - Clinica Dermacross ( Site 0760), Santiago, Region M. de Santiago
  - Espacio Eme ( Site 0762), Santiago, Region M. de Santiago
  - Hospital y CRS El Pino ( Site 0763), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile ( Site 0754), Santiago, Region M. de Santiago
  - Clínica Ensenada ( Site 0753), Santiago, Region M. de Santiago
  - Cardio Sur ( Site 0756), Santiago, Region M. de Santiago
  - Centro De Estudios Cardiologicos Y De Medicina Interna ( Site 0752), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS ( Site 0770), Viña del Mar, Región de Valparaíso
- China (48):
  - Anhui Provincil Hospital South District ( Site 0920), Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University-Cardiovascular ( Site 0856), Beijing, Beijing Municipality
  - Aero Space Center Hospital ( Site 0918), Beijing, Beijing Municipality
  - Beijing Friendship Hospital-Cardology ( Site 0865), Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital ( Site 0911), Beijing, Beijing Municipality
  - The Second Affiliated Hospital Chongqing Medical University-Department of Cardiology ( Site 0908), Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital ( Site 0913), Wanzhou, Chongqing Municipality
  - Lanzhou university second hospital-Lanzhou university second hospital ( Site 0863), Lanzhou, Gansu
  - The First People's Hospital of Foshan ( Site 0898), Foshan, Guangdong
  - Guangdong Provincial People's Hospital-Cardiology ( Site 0852), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Cardiology ( Site 0868), Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University ( Site 0897), Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital-Cardiovascular department ( Site 0895), Shenzhen, Guangdong
  - Hainan General Hospital ( Site 0894), Haikou, Hainan
  - The First Hospital of Harbin Medical University-Cardiology ( Site 0903), Harbin, Heilongjiang
  - Wuhan Union Hospital ( Site 0919), Wuhan, Hubei
  - Changsha Central Hospital ( Site 0854), Changsha, Hunan
  - Hunan Provincial People's Hospital ( Site 0857), Changsha, Hunan
  - Xiangya Hospital Central South University-Cardiological Department ( Site 0899), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University-Cardiology ( Site 0860), Changsha, Hunan
  - BAO TOU CENTRAL HOSPITAL ( Site 0866), Baotou, Inner Mongolia
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Cardiolggy, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Cardiology ( Site 0900), Nanjing, Jiangsu
  - Wuxi No.2 People's Hospital-Cardiology Department ( Site 0877), Wuxi, Jiangsu
  - Wuxi People's Hospital-Cardiovascular Department ( Site 0870), Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 0910), Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital ( Site 0861), Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University-Cardiology Department ( Site 0917), Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Cardiology ( Site 0912), Nanchang, Jiangxi
  - China-Japan Union Hospital-department of cardiology ( Site 0916), Changchun, Jilin
  - Siping Central People's Hospital-Cardiovascular Department ( Site 0915), Siping, Jilin
  - The People's Hospital of Liaoning Province ( Site 0859), Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University ward1 depattment of medical oncology ( Sit, Xi'an, Shaanxi
  - Shaanxi provincial people's hospital ( Site 0853), Xi'an, Shaanxi
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital-Cardiology Department ( Site 0855), Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University-Cardiology ( Site 0851), Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital-Cardiovascular Department ( Site 0905), Shanghai, Shanghai Municipality
  - Shanghai Yangpu District Central Hospital-Cardiology ( Site 0876), Shanghai, Shanghai Municipality
  - Shanghai Xuhui Central Hospital-Cardiovascular Department ( Site 0872), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University ( Site 0904), Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University-Endocrinology ( Site 0902), Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital-Cardiology ( Site 0901), Tianjin, Tianjin Municipality
  - Tianjin People' s Hospital ( Site 0867), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 0907), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine ( Site 0909), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 0914), Hangzhou, Zhejiang
  - People's Hospital of Lishui City-department of cardiovascular ( Site 0862), Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Vasculocardiology Department ( Site 0874, Wenzhou, Zhejiang
- Colombia (12):
  - Fundación Centro de Investigación Clínica CIC ( Site 0955), Medellín, Antioquia
  - Centro Cardiovascular Colombiano Clínica Santa María ( Site 0951), Medellín, Antioquia
  - Rodrigo Botero S.A.S ( Site 0953), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0954), Barranquilla, Atlántico
  - Corazon IPS ( Site 0964), Barranquilla, Atlántico
  - IPS Centro Científico Asistencial S.A.S ( Site 0952), Barranquilla, Atlántico
  - IPS Médicos Internistas de Caldas ( Site 0959), Manizales, Caldas Department
  - Instituto Del Corazón De Bucaramanga ( Site 0960), Bucaramanga, Santander Department
  - Fundación Cardiovascular de Colombia ( Site 0961), Piedecuesta, Santander Department
  - Fundacion Valle del Lili- CIC-Internal Medicine ( Site 0962), Cali, Valle del Cauca Department
  - Centro de Investigaciones Clinicas SAS ( Site 0957), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0963), Cali, Valle del Cauca Department
- Czechia (11):
  - Fakultní nemocnice Brno Bohunice-Interni kardiologicka klinika ( Site 1058), Brno, Brno-mesto
  - Vojenská Nemocnice Brno-Internal department ( Site 1055), Brno, Brno-mesto
  - Nemocnice Slany-Interna - kardiologicka ambulance ( Site 1063), Slaný, Central Bohemia
  - Klinika Dr. Pirka ( Site 1065), Mladá Boleslav, Mlada Boleslav
  - Institut Klinicke a Experimentalni Mediciny-Klinika kardiologie ( Site 1052), Prague, Praha 4
  - Ustredni vojenska nemocnice-Oddeleni kardiologie ( Site 1054), Prague, Praha 6
  - MUDr. Libor Nechvatal s.r.o. , Kardiologie ( Site 1057), Brno, South Moravian
  - Fakultni Nemocnice u sv. Anny v Brne-I. interni kardioangiologicka klinika ( Site 1066), Brno, South Moravian
  - KardioBusak s.r.o. ( Site 1051), Louny
  - Vseobecna fakultni nemocnice v Praze-Centrum srdečního selhání ( Site 1059), Prague
  - KIGE ( Site 1060), Znojmo
- Denmark (13):
  - Rigshospitalet-Cardiology ( Site 1161), Copenhagen, Capital Region
  - Amager Hospital ( Site 1163), Copenhagen, Capital Region
  - Herlev and Gentofte Hospital-Department of Cardiology ( Site 1158), Hellerup, Capital Region
  - Nordsjællands Hospital - Hillerød ( Site 1159), Hillerød, Capital Region
  - Hvidovre Hospital-259 ( Site 1151), Hvidovre, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 1160), Aarhus, Central Jutland
  - Regionshospitalet Viborg ( Site 1166), Viborg, Central Jutland
  - Sygehus Vendsyssel Hjoerring ( Site 1164), Hjørring, North Denmark
  - Holbæk Sygehus-Cardiology ( Site 1152), Holbæk, Region Sjælland
  - Roskilde Sygehus ( Site 1162), Roskilde, Region Sjælland
  - Slagelse Sygehus-Ambulatorium for Hjertesygdomme ( Site 1153), Slagelse, Region Sjælland
  - Sydvestjysk Sygehus Esbjerg-Hjertemedicinsk Projekt ( Site 1154), Esbjerg, Region Syddanmark
  - Svendborg Hospital Odense Universitets hospital-Kardiologisk Forskningsenhed ( Site 1156), Svendborg, Region Syddanmark
- France (11):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur-Service cardiologie ( Site 1353), Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque ( Site 1362), Pessac, Aquitaine
  - Centre Hospitalier Louis Pasteur ( Site 1360), Le Coudray, Eure-et-Loir
  - CHU Rangueil-Cardiology ( Site 1351), Toulouse, Haute-Garonne
  - CHU Charles Nicolle ( Site 1354), Rouen, Haute-Normandie
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitau-Centre Investigation Clinique Plurithé, Vandœuvre-lès-Nancy, Lorraine
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre ( Site 1356), Le Kremlin-Bicêtre, Paris
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer ( Site 1352), Toulon, Provence-Alpes-Côte d'Azur Region
  - Hospices Civils de Lyon - Hopital Louis Pradel ( Site 1364), Lyon, Rhone
  - CHD Vendee ( Site 1361), La Roche-sur-Yon, Vendee
  - Pitie Salpetriere University Hospital ( Site 1363), Paris, Île-de-France Region
- Germany (21):
  - Universitaetsklinikum Heidelberg-Klinik für Kardiologie, Angiologie und Pneumologie ( Site 1475), Heidelberg, Baden-Wurttemberg
  - Klinikum Coburg ( Site 1464), Coburg, Bavaria
  - Kardiologische Gemeinschaftspraxis ( Site 1460), Nuremberg, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 1458), Würzburg, Bavaria
  - ClinPhenomics CVC GmbH ( Site 1457), Frankfurt am Main, Hesse
  - Klinikum Frankfurt Höchst ( Site 1463), Frankfurt am Main, Hesse
  - Asklepios Klinik Langen ( Site 1473), Langen, Hesse
  - Medizinische Hochschule Hannover ( Site 1476), Hanover, Lower Saxony
  - Universitätsmedizin Greifswald ( Site 1470), Greifswald, Mecklenburg-Vorpommern
  - St. Vinzenz-Hospital-Cardiology ( Site 1455), Cologne, North Rhine-Westphalia
  - Klinikum Leverkusen ( Site 1453), Leverkusen, North Rhine-Westphalia
  - Kliniken Maria Hilf-Klinik für Kardiologie ( Site 1454), Mönchengladbach, North Rhine-Westphalia
  - Gemeinschaftspraxis Dr. Fabian Krämer, Dr. Ulrich Overhoff ( Site 1459), Siegen, North Rhine-Westphalia
  - Klinikum Ludwigshafen ( Site 1456), Ludwigshafen am Rhein, Rhineland-Palatinate
  - Marienhaus Klinikum St. Elisabeth Neuwied ( Site 1452), Neuwied, Rhineland-Palatinate
  - Staedtisches Klinikum Dresden-2. Medizinische Klinik ( Site 1468), Dresden, Saxony
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien ( Site 1477), Dresden, Saxony
  - Herzzentrum Dresden GmbH Universitätsklinik ( Site 1469), Dresden, Saxony
  - Katholisches Krankenhaus St. Johann Nepomuk ( Site 1462), Erfurt, Thuringia
  - Praxis Rankestrasse ( Site 1461), Berlin
  - Cardiologicum Hamburg ( Site 1467), Hamburg
- Greece (11):
  - General Hospital of Athens Hippokratio ( Site 1552), Athens, Attica
  - Alexandra Hospital-HEART FAILURE AND CARDIO-ONCOLOGY UNIT ( Site 1559), Athens, Attica
  - General Hospital of Athens "G. Gennimatas"-General Hospital of Athens "G.Gennimatas" ( Site 1561), Athens, Attica
  - Konstantopoulio General Hospital-Cardiology Clinic ( Site 1553), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 1556), Chaïdári, Attica
  - Hygeia Hospital-6th cardiology clinic ( Site 1560), Marousi, Attica
  - University Hospital of Alexandroupolis-First Department of Internal Medicine ( Site 1551), Alexanroupolis, Evros
  - University General Hospital of Larissa ( Site 1555), Larissa, Thessaly
  - University Hospital of Ioannina-2nd Department of Cardiology ( Site 1554), Ioannina, West Greece
  - AHEPA University General Hospital of Thessaloniki-1st Cardiology Clinic ( Site 1558), Thessaloniki
  - European Interbalkan Medical Center-2nd Department of Cardiology ( Site 1557), Thessaloniki
- Guatemala (3):
  - Unidad De Diagnostico Cardiologico ( Site 1652), Guatemala City
  - Clinica Medica ( Site 1651), Guatemala City
  - Unidad De Diagnostico Cardiologico ( Site 1654), Guatemala City
- Hong Kong (4):
  - Grantham Hospital ( Site 1753), Aberdeen
  - Queen Mary Hospital-Medicine - Cardiology ( Site 1752), Hksar
  - Princess Margaret Hospital ( Site 1755), Hong Kong
  - Prince of Wales Hospital ( Site 1751), Shatin
- Hungary (17):
  - CoroMed ( Site 1867), Pécs, Baranya
  - Pécsi Tudományegyetem Klinikai Központ ( Site 1865), Pécs, Baranya
  - Private Practice - Dr. Lakatos Ferenc ( Site 1854), Békéscsaba, Bekes County
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház-Cardiology ( Site 1878), Gyula, Bekes County
  - Bacs-Kiskun Megyei Korhaz-I. Belgyógyászat - Kardiológia ( Site 1873), Kecskemét, Bács-Kiskun county
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Belgyógyászati Klinika ( Site 1874), Szeged, Csongrád megye
  - TaNa Med ( Site 1866), Mosonmagyaróvár, Győr-Moson-Sopron
  - Flor Ferenc Hospital of Pest County-5th Department of Internal Medicine ( Site 1852), Kistarcsa, Pest County
  - CMed Rehabilitacios es Diagnosztikai Kozpont ( Site 1877), Székesfehérvár, Szekesfehervar
  - Tolna Megyei Balassa János Kórház ( Site 1868), Szekszárd, Szekszard
  - DRC Gyógyszervizsgáló Központ ( Site 1869), Balatonfüred, Veszprém megye
  - Szent Rókus Kórház ( Site 1858), Budapest
  - Gottsegen György Országos Kardiovaszkuláris Intézet ( Site 1851), Budapest
  - Semmelweis University-Városmajori Szív- és Érgyógyászati Klinika ( Site 1855), Budapest
  - Óbudai Egészségügyi Centrum ( Site 1861), Budapest
  - Medifarma 98 Kft-Outpatient Clinic ( Site 1859), Nyíregyháza
  - OEC Clinical Research - Zalaegerszeg ( Site 1864), Zalaegerszeg
- Ireland (2):
  - St. Michael's Hospital ( Site 1955), Dún Laoghaire, Dublin
  - St. James's Hospital-Cardiology ( Site 1951), Dublin
- Israel (10):
  - Assuta Ashdod Medical Center-Cardiology ( Site 2063), Ashdod
  - Hillel Yaffe Medical Center-Heart Institute ( Site 2058), Hadera
  - Rambam Health Care Campus-Cardiology ( Site 2053), Haifa
  - Shaare Zedek Medical Center-Cardiology ( Site 2055), Jerusalem
  - Hadassah Medical Center-Heart Institute ( Site 2062), Jerusalem
  - Galilee Medical Center-Cardiology ( Site 2051), Nahariya
  - Rabin Medical Center-Cardiology - CHF ( Site 2052), Petah Tikva
  - Sheba Medical Center-Leviev Heart Center ( Site 2064), Ramat Gan
  - Kaplan Medical Center-Heart Institution ( Site 2054), Rehovot
  - Yitzhak Shamir Medical Center-Cardiology ( Site 2060), Ẕerifin
- Italy (14):
  - Azienda Ospedaliero Universitaria S.Anna ( Site 2152), Cona, Emilia-Romagna
  - Cattinara Hospital-Cardiovascular Department ( Site 2162), Trieste, Friuli Venezia Giulia
  - Policlinico Umberto I ( Site 2166), Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-U.O.C. Cardiologia ( Site 2161), Milan, Lombardy
  - Centro Cardiologico Monzino-Heart Failure Unit ( Site 2153), Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda-Unità Ricerche Cliniche della Cardiologia 4 ( Site 2159), Milan, Milano
  - IRCCS San Raffaele Pisana-riabilitazione cardiologica ( Site 2156), Rome, Roma
  - ospedale le scotte ( Site 2163), Siena, Tuscany
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII-Cardiologia 1 ( Site 2151), Bergamo
  - IRCCS - AOU di Bologna-Dept. of Medical and Surgical sciences ( Site 2158), Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia-Cardiology- Day Hospital ( Site 2154), Brescia
  - Fondazione IRCCS Policlinico San Matteo-Cardiology ( Site 2157), Pavia
  - University of Perugia ( Site 2164), Perugia
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 2165), Torino
- Malaysia (8):
  - Hospital Sultanah Bahiyah-Department of Cardiology ( Site 2355), Alor Star, Kedah
  - Hospital Universiti Sains Malaysia-Medical Department ( Site 2357), Kubang Kerian, Kelantan
  - University Malaya Medical Centre ( Site 2351), Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ( Site 2353), Kuantan, Pahang
  - Hospital Queen Elizabeth II ( Site 2359), Kota Kinabalu, Sabah
  - Sarawak Heart Centre ( Site 2352), Kota Samarahan, Sarawak
  - UiTM Sungai Buloh Campus ( Site 2354), Sungai Buloh, Selangor
  - Hospital Sultanah Nur Zahirah-Jabatan Perubatan ( Site 2360), Kuala Terengganu, Terengganu
- Mexico (23):
  - Medivest Centro de Investigación Integral ( Site 2460), Chihuahua City, Chihuahua
  - CIMAB SA de CV ( Site 2456), Torreón, Coahuila
  - Centro de Investigacion Cardiovascular y Metabólica ( Site 2465), Tijuana, Estado de Baja California
  - Hospital General de Acapulco ( Site 2469), Acapulco de Juárez, Guerrero
  - Grupo Ollin Care ( Site 2476), Pachuca, Hidalgo
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente ( Site 2466), Guadalajara, Jalisco
  - Cardiocent de Guadalajara S.C. ( Site 2464), Guadalajara, Jalisco
  - Instituto Jalisciense de Metabolismo SC ( Site 2467), Guadalajara, Jalisco
  - HOSPITAL GENERAL DE MEXICO DR. EDUARDO LICEAGA ( Site 2478), Mexico City, Mexico City
  - Centro de Imagen y Tecnología en Intervención Cardiovascular ( Site 2477), Mexico City, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez ( Site 2454), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 2474), Mexico City, Mexico City
  - Unidad biomedica avanzada monterrey ( Site 2462), Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral ( Site 2472), San Nicolás de los Garza, Nuevo León
  - Centro de Atención e Investigación Cardiovascular del Potosí ( Site 2453), San Luis Potosí City, San Luis Potosí
  - Centro de Estudios de Alta Especialidad de Sinaloa ( Site 2463), Mazatlán, Sinaloa
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 2468), Ciudad Madero, Tamaulipas
  - Consultorio de Medicina Especilizada del Sector Privado ( Site 2455), Xalapa, Veracruz
  - Hospital Angeles Xalapa ( Site 2451), Xalapa, Veracruz
  - Medical Care and Research SA de CV ( Site 2461), Mérida, Yucatán
  - Fundación Cardiovascular de Aguascalientes A.C. ( Site 2473), Aguascalientes
  - Oaxaca Site Management Organization ( Site 2459), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 2457), Oaxaca City
- New Zealand (7):
  - Christchurch Heart Institute ( Site 2651), Christchurch, Canterbury
  - Dunedin Hospital-Cardiology Department ( Site 2653), Dunedin, Otago
  - Waikato Hospital-Cardiology Clinical Trials Unit ( Site 2654), Hamilton, Waikato Region
  - Hutt Valley District Health board HVDHB-Cardiology Research Unit ( Site 2652), Lower Hutt, Wellington Region
  - North Shore Hospital-Cardiology Research ( Site 2656), Auckland
  - Auckland City Hospital ( Site 2659), Auckland
  - Middlemore Clinical Trials ( Site 2658), Auckland
- Peru (9):
  - Centro de investigacion Clínica Trujillo-Medical specialties ( Site 2860), Trujillo, La Libertad
  - Instituto Nacional Cardiovascular INCOR Carlos Peschiera Carrillo - EsSalud ( Site 2855), Jesús María, Lima
  - Hospital Alberto Sabogal Sologuren ( Site 2851), Bellavista, Qallaw
  - Clínica Vesalio-Cardiology ( Site 2854), Lima
  - Clínica Javier Prado ( Site 2853), Lima
  - Clínica El Golf-Cardiologia ( Site 2857), Lima
  - Clínica Providencia ( Site 2856), Lima
  - Hospital Cayetano Heredia-Servicio de cardiologia ( Site 2852), Lima
  - Clínica Belén ( Site 2858), Piura
- Poland (15):
  - NZOZ Centrum Medyczne KERmed ( Site 3066), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Praktyka Lekarska Lidia Pawlowicz ( Site 3053), Torun, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Zespolony im Ludwika Rydygiera w Toruniu-Oddz.Klin.Kardiologii i Int.T.Kard. ( Si, Torun, Kuyavian-Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca PAKS Małopolskie Centrum Sercowo-Naczyniowe ( Site 3062), Chrzanów, Lesser Poland Voivodeship
  - Centrum Medyczne Zdrowa J. Trebacz, W. Zajdel Sp. J. ( Site 3061), Krakow, Lesser Poland Voivodeship
  - Private Practice - Dr. Robert Witek-Ośrodek Badań Klinicznych "METABOLICA" Lek. Robert Witek ( Site, Tarnów, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski CARDIAMED s.j. ( Site 3070), Legnica, Lower Silesian Voivodeship
  - Instytut Chorób Serca, Zakład Badań Klinicznych Chorób Układu Krążenia ( Site 3057), Wrocaw, Lower Silesian Voivodeship
  - NZOZ Twoja Przychodnia ( Site 3051), Lublin, Lublin Voivodeship
  - SP ZOZ w Puławach- Oddział Kardiologii ( Site 3071), Puławy, Lublin Voivodeship
  - ETG Warszawa ( Site 3052), Warsaw, Masovian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca ( Site 3077), Kędzierzyn-Koźle, Opole Voivodeship
  - Centrum Medyczne Medyk ( Site 3065), Rzeszów, Podkarpackie Voivodeship
  - Centrum Medyczne Dr Sudnik s.c. Wanda i Jerzy Sudnik ( Site 3073), Sokółka, Podlaskie Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii Lek. med. Krzysztof Cymerman, Gdynia, Pomeranian Voivodeship
- Puerto Rico (5):
  - Cooperativa De Facultad Medica Sanacoop-Instituto Sanacoop ( Site 3151), Bayamón
  - Private Practice - Dr. Yolanda Figueroa-Torres ( Site 3156), Humacao
  - Research and Cardiovascular Corp. ( Site 3152), Ponce
  - Caparra Internal Medicine ( Site 3155), Río Grande
  - VA Caribbean Healthcare System ( Site 3157), San Juan
- Russia (19):
  - Ivanovo Regional Healthcare Institution Cardiology Dispensary ( Site 3265), Ivanovo, Ivanovo Oblast
  - Krasnodar Regional Clinical Hospital Number 1 S.V. Ochapovskogo ( Site 3281), Krasnodar, Krasnodarskiy Kray
  - City Hospital No. 4 ( Site 3269), Sochi, Krasnodarskiy Kray
  - First Pavlov State Medical University of Saint Petersburg-Сardiology department ( Site 3257), Saint Petersburg, Leningradskaya Oblast'
  - State budgetary Healthcare Institution of the city of Moscow "V. V. Vinogradov City Clinical Hospita, Moscow, Moscow
  - Omsk Regional Clinical Health Service Number 9 ( Site 3296), Omsk, Omsk Oblast
  - Perm Regional Hospital for War Veterans ( Site 3272), Perm, Permskiy Kray
  - Rostov State Medical University ( Site 3259), Rostov-on-Don, Rostov Oblast
  - Rostov-on-Don City Emergency Hospital ( Site 3271), Rostov-on-Don, Rostov Oblast
  - Ryazan State Medical University named after Academician I.P. Pavlova ( Site 3260), Ryazan, Ryazan Oblast
  - First Pavlov State Medical University of Saint Petersburg ( Site 3288), Saint Petersburg, Sankt-Peterburg
  - Almazov National Medical Research Centre ( Site 3320), Saint Petersburg, Sankt-Peterburg
  - Pokrovskaya Municipal Hospital ( Site 3252), Saint Petersburg, Sankt-Peterburg
  - Pokrovskaya Municipal Hospital-1-st cardiology department ( Site 3251), Saint Petersburg, Sankt-Peterburg
  - Astarta Clinic ( Site 3276), Saint Petersburg, Sankt-Peterburg
  - Clinical Hospital S.R.Mirotvortseva name SSMU ( Site 3254), Saratov, Saratov Oblast
  - Interregional Clinical Diagnostic Center-Department of Clinical Trials ( Site 3307), Kazan', Tatarstan, Respublika
  - Volgograd State Medical University ( Site 3258), Volgograd, Volgograd Oblast
  - Institute for Medical Research ( Site 3316), Saint Petersburg
- Singapore (4):
  - National Heart Centre Singapore ( Site 3351), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 3353), Singapore, Central Singapore
  - Changi General Hospital ( Site 3356), Singapore, South East
  - National University Heart Centre, Singapore-Department of Cardiology ( Site 3355), Singapore, South West
- South Africa (14):
  - Universitas Private Hospital-Cardiology Research ( Site 3453), Bloemfontein, Free State
  - Lenasia Clinical Trial Centre - Johannesburg ( Site 3470), Johannesburg, Gauteng
  - Netcare Sunninghill Hospital ( Site 3457), Johannesburg, Gauteng
  - Midrand Medical Centre ( Site 3466), Midrand, Gauteng
  - University of Pretoria - Faculty of Health Sciences-CRU ( Site 3462), Pretoria, Gauteng
  - Clinical Trial Systems ( Site 3452), Pretoria, Gauteng
  - Jongaie Research ( Site 3469), Pretoria West, Gauteng
  - Chris Hani Baragwanath Academic Hospital ( Site 3455), Soweto, Gauteng
  - Enhancing Care Foundation ( Site 3456), Durban, KwaZulu-Natal
  - Tiervlei Trial Centre ( Site 3461), Bellville, Cape Town, Western Cape
  - TREAD Research ( Site 3451), Cape Town, Western Cape
  - Professor Ntsekhe Cardiology Clinic ( Site 3454), Cape Town, Western Cape
  - Excellentis Clinical Trial Consultants ( Site 3464), George, Western Cape
  - Paarl Research Centre ( Site 3468), Paarl, Western Cape
- South Korea (9):
  - Gachon University Gil Medical Center ( Site 3559), Namdong-gu, Incheon
  - Yonsei University-Wonju Severance Christian Hospital ( Site 3555), Wŏnju, Kang-won-do
  - Chonnam National University Hospital ( Site 3558), Gwangju, Kwangju-Kwangyokshi
  - Hallym University Sacred Heart Hospital-Cardiovascular center ( Site 3556), Anyang-si, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 3551), Cheongju-si, North Chungcheong
  - Pusan National University Hospital-Internal Medicine ( Site 3553), Busan, Pusan-Kwangyokshi
  - Chungnam national university hospital ( Site 3554), Junggu, Taejon-Kwangyokshi
  - Seoul National University Hospital ( Site 3557), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 3552), Seoul
- Spain (12):
  - Hospital Germans Trias i Pujol ( Site 3664), Badalona, Barcelona
  - Hospital Quiron Barcelona ( Site 3655), Barcelona, Catalonia
  - Hospital Universitari de Bellvitge-Unitat Multidisciplinar d'Insuficiència Cardíaca Comunitària (UM, L'Hospitalet de Llobregat, Catalonia
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 3666), A Coruña, La Coruna
  - CHUS - Hospital Clinico Universitario-Cardiology - Clinical Research Unit ( Site 3651), Santiago de Compostela, La Coruna
  - Hospital Universitario Ramón y Cajal ( Site 3662), Madrid, Madrid, Comunidad de
  - HOSPITAL CLINICO DE VALENCIA ( Site 3656), Valencia, Valenciana, Comunitat
  - Parc de Salut Mar - Hospital del Mar ( Site 3663), Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 3659), Barcelona
  - Hospital Clinico San Carlos-Cardiology ( Site 3661), Madrid
  - Hospital Universitario La Paz ( Site 3665), Madrid
  - Hospital Universitario Virgen de Valme ( Site 3654), Seville
- Sweden (9):
  - Falu Lasarett-Dep of Cardiology ( Site 3756), Falun, Dalarna County
  - Clemenstorgets Hjartmottagning ( Site 3755), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna-Heart and Vascular theme ( Site 3759), Solna, Stockholm County
  - Aleris Specialistvård Sabbatsberg ( Site 3762), Stockholm, Stockholm County
  - Akardo Med Site ( Site 3763), Stockholm, Stockholm County
  - Skellefteå Lasarett-Research unit, floor 5 ( Site 3760), Skellefteå, Västerbotten County
  - Västmanlands Sjukhus Västerås ( Site 3757), Västerås, Västmanland County
  - Sahlgrenska Universitetssjukhuset-Cardiology Research Unit ( Site 3753), Gothenburg, Västra Götaland County
  - Universitetssjukhuset Örebro-Heart-Lung-Physiology Clinic ( Site 3754), Örebro, Örebro County
- Taiwan (6):
  - Changhua Christian Hospital ( Site 3857), Changhua County, Changhua
  - Mackay Memorial Hospital-Hsinchu ( Site 3852), Hsinchu, Hsinchu
  - Kaohsiung Medical University Hospital ( Site 3856), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 3855), Taichung
  - Taipei Veterans General Hospital-General Clinical Research Center ( Site 3851), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3854), Taoyuan District
- Turkey (Türkiye) (13):
  - Ege University Medicine of Faculty-Cardilogy Department ( Site 4054), Bornova, İzmir
  - Afyon Kocatepe Üniversitesi Tıp Fakültesi-Cardiology Department ( Site 4058), Afyonkarahisar
  - Hacettepe Universitesi ( Site 4061), Ankara
  - Ankara Bilkent Şehir Hastanesi-cardiology ( Site 4053), Ankara
  - Antalya Egitim ve Arastırma Hastanesi-Cardiology ( Site 4064), Antalya
  - Eskisehir Osmangazi University-Cardiology ( Site 4052), Eskişehir
  - Istanbul University Cerrahpasa Medical School Internal Diseases Institute-CARDIOLOGY INSTITUTE ( Sit, Istanbul
  - Başkent Üniversitesi Istanbul Hastanesi ( Site 4057), Istanbul
  - Dr. Siyami Ersek Göğüs Kalp Ve Damar Cerrahisi Eğitim Ve Araştırma Hastanesi ( Site 4063), Istanbul
  - Dokuz Eylül Üniversitesi-CARDIOLOGY ( Site 4055), Izmir
  - Medical Park zmir Hastanesi-cardiology ( Site 4059), Izmir
  - Kocaeli Üniversitesi-Cardiology ( Site 4060), Kocaeli
  - Mersin University ( Site 4056), Mersin
- Ukraine (24):
  - Communal non-profit enterprise "Cherkasy Regional Hospital of Сherkasy Regional Council" ( Site 4292, Cherkasy, Cherkasy Oblast
  - Cherkasy Regional Hospital-Cardiorheumatology ( Site 4283), Cherkasy, Cherkasy Oblast
  - Clinical medical and diagnostic center Limited Liability Company "Simedgroup" ( Site 4284), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Municipal Non-commercial Enterprise "Ivano-Frankivsk Regional Clinical Cardiology Center of Ivano-Fr, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Central clinical hospital - Ukrzalisnytsia-2nd Cardiology ( Site 4306), Kharkiv, Kharkivs’ka Oblast’
  - Communal non-profit enterprise "City Clinical Hospital # 27" of Kharkiv City Council ( Site 4262), Kharkiv, Kharkivs’ka Oblast’
  - L.T. Mala National Institute of Therapy of NAMS of Ukraine-Clinical Pharmacology and Pharmacogeneti, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-Profit Enterprise -City clinical hospital No8 of Kharkiv city council ( Site 4278), Kharkiv, Kharkivs’ka Oblast’
  - Khmelnytskyi Regional Cardiovascular Center-department of invasive cardiology and interventional ra, Khmelnytskyi, Khmelnytskyi Oblast
  - Kyiv Railway Clinical Hospital No.2 of Branch Health Center of the Public Joint Stock Company Ukrain, Kiev, Kyiv Oblast
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical" ( Site 4257), Kiev, Kyiv Oblast
  - Medbud Clinic ( Site 4265), Kyiv, Kyivska Oblast
  - State Institution National Scientific Center M.D. Strazhesko-Essential Hypertension ( Site 4259), Kyiv, Kyivska Oblast
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council ( Site 42, Odesa, Odesa Oblast
  - Ukrayins'kyy Derzhavnyy Naukovo-Doslidnyy Instytut Rebilitatsiyi Invalidiv ( Site 4274), Vinnytsia, Vinnytsia Oblast
  - Lutsk City Clinical Hospital-Center for Cardiovascular Disease ( Site 4255), Lutsk, Volyn Oblast
  - Zakarpattya Regional Clinical Cardiology Dispensary-Dept. of Hospital Therapy, Uzhhorod National Un, Uzhhorod, Zakarpattia Oblast
  - Communal Non-profit Enterprise "City Hospital #6" Zaporizhzhia City Counci-Therapy department ( Site, Zaporizhia, Zaporizhzhia Oblast
  - Communal nonprofit enterprise "City Hospital #9" of Zaporizhzhia City Council ( Site 4251), Zaporizhia, Zaporizhzhia Oblast
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council-Advisory and Treatment department of Sci, Zhytomyr, Zhytomyr Oblast
  - Consultative - Diagnostic Centre of Pechersky District-Therapeutic department ( Site 4307), Kyiv
  - MNE " Kyiv City Clinical Emergency Hospital" of Kyiv Regional Council (KCSA) ( Site 4256), Kyiv
  - State Institution National Scientific Center M.D. Strazhesko-Department of clinical arrhythmology a, Kyiv
  - State Institution National Scientific Center M.D. Strazhesko-Resuscitation and Intensive care ( Site, Kyiv
- United Kingdom (20):
  - Cumberland Infirmary ( Site 4174), Carlisle, Cumbria
  - West Cumberland Hospital ( Site 4176), Whitehaven, Cumbria
  - Chesterfield Royal Hospital ( Site 4159), Calow Chesterfield, Derbyshire
  - Ninewells Hospital and Medical School-Cardiology ( Site 4164), Dundee, Dundee City
  - Carmel Medical Practice ( Site 4152), Darlington, England
  - Russells Hall Hospital ( Site 4153), Dudley, England
  - King's College Hospital-Cardiac Research Department ( Site 4154), London, England
  - St. George's Hospital-Cardiology Clinical Academic Group ( Site 4156), London, England
  - Prince Charles Hospital ( Site 4171), Merthyr Tydfil, Great Britain
  - Layton Medical Centre ( Site 4184), Blackpool, Lancashire
  - Ulster Hospital ( Site 4185), Belfast, Lisburn And Castlereagh
  - William Harvey Heart Centre ( Site 4169), London, London, City of
  - Craigavon Area Hospital ( Site 4162), Belfast, Northern Ireland
  - Princess of Wales Hospital ( Site 4178), Bridgend, Wales
  - Walsall Manor Hospital ( Site 4179), West Midlands, Walsall
  - Worcestershire Royal Hospital-Cardiology Research Department ( Site 4181), Worcester, Worcestershire
  - Blackpool Victoria Hospital ( Site 4161), Blackpool
  - University Hospital Coventry & Warwickshire-Research & Development ( Site 4170), Coventry
  - The Adam Practice ( Site 4180), Poole
  - University Hospital of North Tees ( Site 4172), Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Butler J, Usman MS, Anstrom KJ, Blaustein RO, Bonaca MP, Ezekowitz JA, Freitas C, Lam CSP, Lewis EF, Lindenfeld J, McMullan CJ, Mentz RJ, O'Connor C, Rosano GMC, Saldarriaga CI, Senni M, Udelson J, Voors AA, Zannad F. Soluble guanylate cyclase stimulators in patients with heart failure with reduced ejection fraction across the risk spectrum. Eur J Heart Fail. 2022 Nov;24(11):2029-2036. doi: 10.1002/ejhf.2720. Epub 2022 Nov 16. PMID 36250238
- [Result] Reddy YNV, Butler J, Anstrom KJ, Blaustein RO, Bonaca MP, Corda S, Ezekowitz JA, Lam CSP, Lewis EF, Lindenfeld J, McMullan CJ, Mentz RJ, O'Connor C, Patel M, Ponikowski P, Rosano GMC, Saldarriaga CI, Senni M, Udelson J, Voors AA, Zannad F. Vericiguat Global Study in Participants with Chronic Heart Failure: Design of the VICTOR trial. Eur J Heart Fail. 2025 Feb;27(2):209-218. doi: 10.1002/ejhf.3501. Epub 2024 Oct 30. PMID 39473305
- [Result] Butler J, McMullan CJ, Anstrom KJ, Barash I, Bonaca MP, Borentain M, Corda S, Ezekowitz JA, Felker GM, Gates D, Lam CSP, Lewis EF, Lindenfeld J, Mentz RJ, O'Connor CM, Ponikowski P, Reddy YNV, Rosano GMC, Saldarriaga C, Senni M, She L, Teixeira PP, Udelson J, Urbinati A, Vlajnic V, Voors AA, Xing A, Patel MJ, Zannad F; VICTOR Study Group. Vericiguat in patients with chronic heart failure and reduced ejection fraction (VICTOR): a double-blind, placebo-controlled, randomised, phase 3 trial. Lancet. 2025 Sep 27;406(10510):1341-1350. doi: 10.1016/S0140-6736(25)01665-4. Epub 2025 Aug 30. PMID 40897189
- [Derived] Khan MS, Grayburn PA, Butler J. Cardiac reverse remodelling with vericiguat: Victory or no victory? Eur J Heart Fail. 2023 Jul;25(7):1022-1024. doi: 10.1002/ejhf.2883. Epub 2023 May 25. No abstract available. PMID 37191077
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26239&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 10923 participants screened, 6106 participants were randomized in a 1:1 ratio to receive either vericiguat or matching placebo.
  One participant was randomized in the study at 2 different clinical study sites. Due to double enrolment and study site noncompliance with Good Clinical Practice (GCP), this participant was excluded from all efficacy and safety analyses. Results are presented based on 6105 randomized participants.
Groups:
- Vericiguat: Participants received a starting dose of 2.5 mg of vericiguat taken orally once daily for 2 weeks. The vericiguat dose was titrated to 5 mg for 2 weeks and then to the target dose of 10 mg for the remainder of treatment (total treatment of up to approximately 37 months).
- Placebo: Participants received a placebo matched to the vericiguat dose of 2.5 mg taken orally once daily for 2 weeks. The placebo dose was sham titrated to 5 mg for 2 weeks and then to 10 mg for the remainder of treatment (total treatment of up to approximately 37 months).
Period: Overall Study
Arm/Group | Vericiguat | Placebo
Started | 3053 | 3052
Treated | 3049 | 3049
Completed | 2648 | 2571
Not Completed | 405 | 481
Not completed — Death | 372 | 434
Not completed — Lost to Follow-up | 13 | 16
Not completed — Physician Decision | 0 | 2
Not completed — Sponsor Decision | 1 | 3
Not completed — Withdrawal by Guardian | 1 | 1
Not completed — Withdrawal by Subject | 18 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vericiguat | Placebo | Total
Number analyzed (Participants) | 3053 | 3052 | 6105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (11.0) | 67.0 (11.0) | 67.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 727 | 713 | 1440
  Male | 2326 | 2339 | 4665
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 968 | 953 | 1921
  Not Hispanic or Latino | 2044 | 2068 | 4112
  Unknown or Not Reported | 41 | 31 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 159 | 142 | 301
  Asian | 383 | 363 | 746
  Native Hawaiian or Other Pacific Islander | 4 | 7 | 11
  Black or African American | 251 | 218 | 469
  White | 1942 | 1992 | 3934
  More than one race | 313 | 330 | 643
  Unknown or Not Reported | 1 | 0 | 1
New York Heart Association (NYHA) Functional Classification (FC) of Heart Failure [Count of Participants; unit: Participants] — Participants were stratified by: NYHA FC II versus NYHA FC III/IV. Participants were assessed for 1 of 4 NYHA functional classes based on symptoms: Class I (No limitation of physical activity [PA]); Class II (Slight limitation of PA, comfortable at rest, ordinary PA causes fatigue, palpitation, dyspnea, or anginal pain); Class III (Marked limitation of PA, comfortable at rest, less-than-ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain); Class IV (Unable to carry on any PA without discomfort, symptoms of heart failure at rest).
  Participants
    NYHA Class II | 2411 | 2411 | 4822
    NYHA Class III/IV | 642 | 641 | 1283

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Composite Endpoint of Cardiovascular (CV) Death or Heart Failure (HF) Hospitalization: Participants With an Event Per 100 Patient-Years
Description: The time to first occurrence of the composite endpoint of CV death or HF hospitalization was defined as the time from randomization to the first event of CV death or HF hospitalization. Randomized participants without a HF hospitalization or CV death event at the time of analysis were censored at the last available information, when the protocol pre-specified number of total CV death events was achieved (primary completion analysis data cutoff), or the date of their non-CV death, whichever occurred first. Events were confirmed by a clinical events committee (CEC). Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of participants with a CV death or HF hospitalization event per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Pts. with event/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Pts. with event/100 patient-yrs at risk | 11.3 | 12.2
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.219, Log Rank; Stratified by the randomization stratification factor (NYHA FC); Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.83 to 1.04] — Based on a Cox proportional hazard model controlling for the randomization stratification factor (NYHA FC)

2. Secondary Outcome: Time to CV Death: Participants With an Event Per 100 Patient-Years
Description: Time to CV death was defined as the time from randomization to CV death. Randomized participants without a CV death at the time of analysis were censored at their last available information, when the protocol pre-specified number of total CV death events was achieved (primary analysis database cutoff), or the date of their non-CV death, whichever occurred first. CV deaths were confirmed by a CEC. Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of participants with a CV death event per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Pts. with event/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Pts. with event/100 patient-yrs at risk | 5.7 | 6.8
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.020, Log Rank; Stratified by the randomization stratification factor (NYHA FC); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.71 to 0.97] — Based on a Cox proportional hazard model controlling for the randomization stratification factor (NYHA FC)

3. Secondary Outcome: Time to First Occurrence of HF Hospitalization: Participants With an Event Per 100 Patient-Years
Description: Time to first occurrence of HF hospitalization was defined as the time from randomization to the first event of HF hospitalization. Randomized participants without an HF hospitalization at the time of analysis were censored at their last available information, when the protocol pre-specified number of total CV death events was achieved (primary analysis database cutoff), or the date of their death, whichever occurred first. HF hospitalizations were confirmed by a CEC. Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of participants with an HF hospitalization event per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Pts. with event/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Pts. with event/100 patient-yrs at risk | 7.2 | 7.6
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.509, Log Rank; Stratified by the randomization stratification factor (NYHA FC); Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.82 to 1.10] — Based on a Cox proportional hazard model controlling for the randomization stratification factor (NYHA FC)

4. Secondary Outcome: Time to Total HF Hospitalizations (Including First and Recurrent Events): Total Events Per 100 Patient-Years
Description: Time to total HF hospitalizations was defined as the time from randomization to all HF hospitalization events, including time to first event and time increments between events. Randomized participants without an HF hospitalization at the time of analysis were censored at their last available information, when the protocol pre-specified number of total CV death events was achieved (primary analysis database cutoff), or the date of their death, whichever occurred first. HF hospitalizations were confirmed by a CEC. Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of total HF hospitalization events per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Total events/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Total events/100 patient-yrs at risk | 10.7 | 11.8
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.094, Andersen-Gill Model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.80 to 1.02] — Based on an Andersen-Gill model controlling for the randomization stratification factor (NYHA FC)

5. Secondary Outcome: Time to First Occurrence of Composite Endpoint of All-Cause Mortality or HF Hospitalization: Participants With an Event Per 100 Patient-Years
Description: The time to first occurrence of the composite endpoint of all-cause mortality or HF hospitalization was defined as the time from randomization to the first event of all-cause mortality or HF hospitalization. Randomized participants without an all-cause mortality or HF hospitalization event at the time of analysis were censored at the last available information or when the protocol pre-specified number of total CV death events is achieved (primary analysis database cutoff), whichever occurred first. Events were confirmed by a CEC. Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of participants with an all-cause mortality or HF hospitalization event per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Pts. with event/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Pts. with event/100 patient-yrs at risk | 12.7 | 13.9
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.116, Log Rank; Stratified by the randomization stratification factor (NYHA FC); Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.82 to 1.02] — Based on a Cox proportional hazard model controlling for the randomization stratification factor (NYHA FC)

6. Secondary Outcome: Time to All-Cause Mortality: Participants With an Event Per 100 Patient-Years
Description: Time to all-cause mortality was defined as the time from randomization to all-cause mortality. Randomized participants without an all-cause mortality event at the time of analysis were censored at their last available information or when the protocol pre-specified number of total CV death events was achieved (primary analysis database cutoff), whichever occurred first. All-cause mortality was confirmed by a CEC. Protocol-specified final analyses are reported here with a primary completion data cutoff. Time-to-event methodology was used to evaluate the results and the number of participants with an all-cause mortality event per 100 patient-years at risk is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who had GCP-compliant data collected.
Measure: Number; unit: Pts. with event/100 patient-yrs at risk
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3053 | 3052
Pts. with event/100 patient-yrs at risk | 7.3 | 8.6
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Superiority; p = 0.015, Log Rank; Stratified by the randomization stratification factor (NYHA FC); Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.74 to 0.97] — Based on a Cox proportional hazard model controlling for the randomization stratification factor (NYHA FC)

7. Secondary Outcome: Percentage of Participants Who Experienced One or More Selected Nonserious Adverse Events (NSAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Selected NSAEs are defined as nonserious AEs that meet any of the following criteria: AEs that lead to study intervention dose modification or discontinuation, AEs that lead to withdrawal from the study, or Coronavirus Disease 2019 (COVID-19) disease-related AEs. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more selected NSAEs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of participants | 19.7 | 16.9

8. Secondary Outcome: Percentage of Participants Who Experienced One or More Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or other important medical events as determined by the investigator. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more SAEs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of participants | 23.5 | 24.6

9. Secondary Outcome: Percentage of Participants Who Experienced One or More Events of Clinical Interest (ECIs)
Description: ECIs were determined and reported based on the clinical judgment of the investigator. As pre-specified in the protocol, ECIs included the following: 1) Events of potential drug-induced liver injury (DILI), defined as an elevated aspartate aminotransferase or alanine aminotransferase laboratory value that is greater than or equal to 3X the upper limit of normal (ULN) and an elevated total bilirubin laboratory value that is greater than or equal to 2X the ULN and, at the same time, an alkaline phosphatase laboratory value that is less than 2X the ULN, 2) Events associated with symptomatic hypotension, or 3) Events associated with anemia, regardless of etiology. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more ECIs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of participants | 17.6 | 14.6

10. Secondary Outcome: Percentage of Participants Who Experienced One or More Potential DILI ECIs
Description: Potential DILI ECIs were determined and reported based on the clinical judgment of the investigator. Potential DILI ECIs were defined as an elevated aspartate aminotransferase or alanine aminotransferase laboratory value that is greater than or equal to 3X the ULN and an elevated total bilirubin laboratory value that is greater than or equal to 2X the ULN and, at the same time, an alkaline phosphatase laboratory value that is less than 2X the ULN. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more potential DILI ECIs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of Participants | 0.3 | 0.4
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other; p = 0.512, Miettinen and Nurminen; Difference in Percentage = -0.1, 95% CI 2-sided [-0.4 to 0.2]

11. Secondary Outcome: Percentage of Participants Who Experienced One or More Symptomatic Hypotension ECIs
Description: Symptomatic hypotension ECIs were determined and reported based on the clinical judgment of the investigator. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more symptomatic hypotension ECIs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of Participants | 11.3 | 9.2
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other; p = 0.007, Miettinen and Nurminen; Difference in Percentage = 2.1, 95% CI 2-sided [0.6 to 3.6]

12. Secondary Outcome: Percentage of Participants Who Experienced One or More Anemia ECIs
Description: Anemia ECIs were determined and reported based on the clinical judgment of the investigator, regardless of etiology. Protocol-specified final analyses are reported here with a primary completion data cutoff. The percentage of participants who experienced one or more anemia ECIs is presented.
Time Frame: Up to approximately 36 months (from randomization to the primary completion data cutoff)
Population: All randomized participants who received at least 1 dose of study intervention and who had GCP-compliant data collected.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 3049 | 3049
Percentage of Participants | 7.6 | 6.3
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other; p = 0.045, Miettinen and Nurminen; Difference in Percentage = 1.3, 95% CI 2-sided [0.0 to 2.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 39 months (duration over which AEs were monitored at the participant level; from randomization to study completion data cutoff)
Description: One participant was enrolled at 2 study sites and was excluded from all analyses due to GCP-noncompliant data. All-Cause Mortality: all randomized participants. SAEs and Other AEs: all participants who received ≥1 dose of study intervention. All SAEs were reported. As pre-specified in the protocol, only selected Other AEs were reported, related to potential DILI, hypotension, anemia, COVID-19-related AEs, and AEs causing study discontinuation or study drug dose modification or discontinuation.
Arm/Group | Vericiguat | Placebo
All-Cause Mortality (participants affected / at risk) | 392/3053 | 455/3052
Serious Adverse Events (participants affected / at risk) | 732/3049 | 766/3049
Other Adverse Events (participants affected / at risk) | 530/3049 | 423/3049
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=3049) | Placebo (N=3049)
Anaemia (Blood and lymphatic system disorders) | 26 (28) | 34 (35)
Anaemia macrocytic (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 5 (6)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 14 (15)
Angina pectoris (Cardiac disorders) | 5 (5) | 4 (4)
Angina unstable (Cardiac disorders) | 4 (4) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmic storm (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 24 (26) | 24 (26)
Atrial flutter (Cardiac disorders) | 2 (2) | 4 (4)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (5) | 3 (3)
Cardiac failure (Cardiac disorders) | 122 (134) | 117 (136)
Cardiac failure acute (Cardiac disorders) | 9 (11) | 14 (17)
Cardiac failure chronic (Cardiac disorders) | 12 (13) | 7 (7)
Cardiac failure congestive (Cardiac disorders) | 10 (10) | 12 (12)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 10 (10) | 16 (16)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Cardiorenal syndrome (Cardiac disorders) | 4 (4) | 3 (4)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 11 (11) | 10 (12)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (2)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure with reduced ejection fraction (Cardiac disorders) | 0 (0) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 9 (9) | 3 (3)
Myocardial infarction (Cardiac disorders) | 9 (9) | 8 (8)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 4 (4)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 5 (6) | 7 (7)
Ventricular flutter (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 14 (16) | 22 (25)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Reproductive tract hypoplasia, male (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Primary adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 6 (6)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 12 (12)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 7 (7)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric arteriosclerosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 5 (5) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (9) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 4 (4)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (5) | 5 (5)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Medical device site haematoma (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 6 (6) | 6 (6)
Non-cardiac chest pain (General disorders) | 7 (8) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 3 (3)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Suspected drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 2 (3) | 0 (0)
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Biliary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 7 (7) | 5 (5)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 20 (20) | 24 (24)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 9 (9) | 15 (16)
Chagas' cardiomyopathy (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 5 (5)
Device related infection (Infections and infestations) | 2 (2) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 2 (2)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 3 (3)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 4 (4)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Endotoxaemia (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 11 (11) | 8 (9)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 4 (4)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 4 (5)
Influenza (Infections and infestations) | 5 (5) | 5 (5)
Intervertebral discitis (Infections and infestations) | 0 (0) | 2 (2)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 8 (8) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3) | 4 (5)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 73 (83) | 78 (88)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 7 (9) | 6 (6)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 2 (2)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 14 (14) | 18 (18)
Septic shock (Infections and infestations) | 12 (12) | 19 (19)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 19 (19) | 17 (18)
Urosepsis (Infections and infestations) | 6 (6) | 6 (6)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 4 (4) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 9 (9)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 7 (7)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 2 (3)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 3 (3) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 2 (2)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (7) | 14 (15)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant nipple neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome with single lineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 4 (4)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 3 (3)
Dementia (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 2 (2)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Miller Fisher syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 3 (3)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 18 (19) | 13 (13)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 3 (3)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 3 (3) | 2 (2)
Device power source issue (Product Issues) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1) | 1 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 32 (32) | 56 (62)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 15 (17) | 16 (18)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (4) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 17 (18) | 7 (7)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 6 (6)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 5 (6) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (27) | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 2 (2)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Distributive shock (Vascular disorders) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive end-organ damage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 30 (32) | 29 (29)
Hypovolaemic shock (Vascular disorders) | 3 (3) | 2 (2)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 12 (12)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular haematoma (Vascular disorders) | 1 (1) | 0 (0)
Scalp haematoma (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=3049) | Placebo (N=3049)
Anaemia (Blood and lymphatic system disorders) | 171 (190) | 143 (154)
Hypotension (Vascular disorders) | 401 (502) | 312 (380)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05093933/Prot_SAP_000.pdf